CLINICAL TRIAL: NCT06189768
Title: A Retrospective Study on Pigmentation Disorders in Children in a Tertiary Care Children's Hospital.
Brief Title: A Study on Pigmentation Disorders in Children
Status: Completed | Type: Observational
Sponsor: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Abal Baral, Principal Investigator, Nepal Health Research Council
Other Study IDs: 59/2020-021
Record Dates: First submitted 2023-12-13; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Hyperpigmentation; Pediatric Dermatology
Keywords: Hyperpigmentation disorders; Nepal; Pediatric; Observational study
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with hyperpigmentation disorder: Children aged 0 to 15 with hyperpigmentation due to any cause presenting to Dermatology Outpatient Department of Kanti Children's Hospital

SUMMARY:
The descriptive cross-sectional study was undertaken at Kanti Children's Hospital during the period from January 2020 to June 2021. Ethical approval for the study was obtained from the Institutional Review Board of Kanti Children's Hospital (IRB-KCH). The refence number is 59/2020-021. The study focused on children with hyperpigmentation disorders presenting at the Dermatology Outpatient Department of Kanti Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* children ranging from newborns to 15 years old with hyperpigmentation due to any cause

Exclusion Criteria:

* children admitted to wards

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Inclusive of children ranging from newborns to 15 years old with hyperpigmentation due to any cause, the study excluded those admitted to wards with alternative diagnoses.
Study Population: Inclusive of children ranging from newborns to 15 years old with hyperpigmentation due to any cause, the study excluded those admitted to wards with alternative diagnoses
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Measure the causes of hyperpigmentation in children aged 0 to 15 | 1.5 years
  Measure the prevalence of different causes of hyperpigmentation due to any cause in children aged 0 to 15 years presenting to the dermatology outpatient department of Kanti Children's Hospital. Outpatient hospital records were used for collecting the study variables.
Measure the age distribution of children with hyperpigmentation disorders | 1.5 years
  The age (in years) of all the children with hyperpigmentation disorders presenting to the outpatient department of Kanti Children's Hospital was recorded. Outpatient hospital records were used for collecting the study variable.
Measure the gender distribution of children with hyperpigmentation disorders | 1.5 years
  The gender (male or female) of all the children with hyperpigmentation disorders presenting to the outpatient department of Kanti Children's Hospital was recorded. Outpatient hospital records were used for collecting the study variable.
Measure the caste distribution of children with hyperpigmentation disorders | 1.5 years
  The caste of all the children with hyperpigmentation disorders presenting to the outpatient department of Kanti Children's Hospital was recorded. Outpatient hospital records were used for collecting the study variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanti Children's Hospital, Kathmandu, Nepal